CLINICAL TRIAL: NCT00677404
Title: Evaluation of Clinical Outcome in Advanced Chronic Lower Limb Ischemia by Stem Cell Transplantation With or Without (Granulocyte-colony Stimulation Factor) G-CSF Injection
Brief Title: Autologous Transplantation of Bone Marrow Mononuclear Cell (BM-MNC) With and Without Granulocyte-Colony Stimulation Factor (G-CSF) for Treatment of Chronic Lower Limb Ischemic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Hamid Gourabi, Chief, Royan Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-PVD-001
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2010-04

CONDITIONS: Peripheral Vascular Diseases; Ischemia
Keywords: Peripheral vascular diseases; chronic lower limb ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stem cell recipient (Experimental): the patients with peripheral vascular disease who receive bone marrow derived mono nuclear cells
  Interventions: Biological: BM-MNC injection

INTERVENTIONS:
Biological: BM-MNC injection — Bone marrow aspiration A total volume of 400 ml bone marrow will be aspirated from the iliac crest under epidural anaesthesia

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of mononuclear cells with and without G-CSF in patients with chronic lower limb ischemia.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) results from severe occlusive disease that impairs distal limb perfusion to the point where oxygen delivery is no longer adequate to meet the metabolic needs of the tissue, even under resting conditions. The limits of peripheral artery disease (PAD) compensatory mechanisms, such as distal vasodilatation and collateral formation, have been exceeded at this point. PAD is a widespread disease, affecting up to 15% of all adults older than 55 years. Formation of true new blood vessels, or angiogenesis, and development of collateral vessels from preexisting blood vessels, or arteriogenesis, is important in the pathophysiology of vascular disease. By stimulating these processes we might be able to provide an alternative treatment strategy for patients with lower limb ischemia. In response to tissue injury and remodeling, neovascularization usually occurs via the proliferation and migration of progenitor endothelial cells (EPC) from preexisting vasculature. The EPCs resident within bone marrow and peripheral blood, so it seems implantation of BM cells can contribute to injury-induced and pathology induced neovascularization. Indeed, recent studies have shown that bone-marrow mononuclear cell (BM-MNC) implantation increases collateral vessel formation in both ischemic limb models and patients with limb ischemia. In addition, granulocyte-colony stimulation factor could mobilize the EPCs to peripheral blood. After BM-MNC implantation, G-CSF can contribute more EPC in PB for effective angiogenesis in PAD patients.

In this study, Bone marrow puncture will be performed in a common manner. The iliac crest is punctured under epidural anesthesia and 400 mL of bone marrow will be aspirated. The MNCs are isolated under good manufacturing practice conditions by Ficoll density separation and is intramuscularly injected (40 sites, in 3 × 3 cm distance, 1-1.5 cm deep, into ischemic leg. In some patients G-CSF (10 microgr/day) is administration by subcutaneous injection from day of cell injection for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Critical Limb ischemia according to the guidelines of the Transatlantic Consensus Group (TASC) Rutherford grade II or III. Perfusion is measured with absolute perfusion pressure and ankle-brachial index (ABI) and transcutaneous oxygen tension (TcpO2); for inclusion, ABI has to be less than or equal to 0.6 or absolute ankle pressure must be less than 60 mmHg. If ABI is technically not feasible, e.g. in patients with media calcification, inclusion criteria are a tcpO2 value (supine, forefoot, 44°C) of less than 20 mmHg if there is no tissue loss, or a tcpO2 of less than 40 mmHg if there is tissue loss.
* No sufficient response to best standard care delivered for six weeks.
* No surgical or radiological interventional option for revascularisation as confirmed by a vascular surgeon and an interventional radiologist
* Signed informed consent
* Absence of life-threatening complications from the ischemic limb

Exclusion Criteria:

* Expected life span less than six months
* Bone marrow diseases which preclude transplantation (eg lymphoma, leukaemia, myelodysplastic syndrome and others)
* Patients with poorly controlled diabetes mellitus (HbA1C > 8%)
* Patients with renal insufficiency (creatinine > 2.5).
* Patients with evidence of infectious disease as determined by e. above or other medical findings.
* Pregnant women (women capable of childbearing must have a negative pregnancy test).
* Patients with cognitive impairments.
* Other comorbid disease that would be expected to result in less than one year life expectancy
* Past malignancy or history of chemotherapy or radiation affecting the bone marrow.
* History of inflammatory or progressively fibrotic conditions: .e.g., rheumatoid arthritis, systemic lupus erythematosis, vasculitic disorders, idiopathic pulmonary fibrosis, retroperitoneal fibrosis
* Infection as evidenced by WBC count of >15,000 and/or temperature more than 38C. Large area of cellulitis in the afflicted limb that in the opinion ofthe investigators would require the institution of antibiotics OR evidence of osteomyelitis corroborated by radiographic or scintigraphic examination
* Cardiovascular conditions:
* EF<30%
* Acute ST elevation myocardial infarction (MI) within 1month;
* Transient ischemic attack or stroke within 1 month;
* Severe valvular disease
* CVA
* Patients with any history of organ transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Major amputation | six months

SECONDARY OUTCOMES:
Minor amputation | six months
Number and extent of leg ulcers | six months
Resolvement of rest pain | six months
Improvement of ankle-brachial index (ABI) | six months
Improvement of pain free walking distances ( PFWD) | six months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gorabi, PhD, Study Chair — Royan institute, Tehran, Iran; Mohammad reza Zafarghandi, MD, Study Chair — Sina Hospital, Tehran, Iran; Nasser Aghdami, MD., PhD, Study Director — Royan institute, Tehran, Iran; Hossein Baharvand, PhD, Principal Investigator — Royan institute, Tehran, Iran; Hassan Ravari, MD, Principal Investigator — Sina Hospital, Tehran, Iran
Locations (2):
- Iran (2):
  - Royan Institute, Tehran, Tehran Province
  - Tehran University of medical sciences, Vascular Surgery department, Sina Hospital, Tehran, Tehran Province

REFERENCES:
- [Result] Zafarghandi MR, Ravari H, Aghdami N, Namiri M, Moazzami K, Taghiabadi E, Fazel A, Pournasr B, Farrokhi A, Sharifian RA, Salimi J, Moini M, Baharvand H. Safety and efficacy of granulocyte-colony-stimulating factor administration following autologous intramuscular implantation of bone marrow mononuclear cells: a randomized controlled trial in patients with advanced lower limb ischemia. Cytotherapy. 2010 Oct;12(6):783-91. doi: 10.3109/14653240903518163. PMID 20078390
- See also: Related Info — http://www.royaninstitute.org